CLINICAL TRIAL: NCT05431465
Title: Evaluation of Wear Behavior of Onlay Restorations Constructed From Two Types of Glass Ceramics
Brief Title: Wear of Vita Ambria Only Restoration Compared With IPS Emax Onlay Restoration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Abd Elaziz Helmy Abd Elaziz Mahmoud Elhamrawy, Assistant lecturer, Department of Crown&Bridge,Al-Azhar Unverisity, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Wear of Vita Ambria
Record Dates: First submitted 2022-06-20; First posted 2022-06-24 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Carious Tooth; Dental Wear
MeSH Terms: conditions — Tooth Wear

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vita Ambria onlay (Experimental): The onlays will be constructed from Zirconia reinforced Lithium disilicate (Vita Ambria) glass ceramic system.
  Interventions: Other: Vita Ambria
- IPS emax onlay (Active Comparator): The onlays will be constructed from Lithium disilicate (IPS e-max press) glass ceramic system
  Interventions: Other: IPs emax onaly

INTERVENTIONS:
Other: Vita Ambria — onlay restoration will be fabricated from Zirconia reinforced lithium disilicate glass ceramic(vita ambria)
  Arms: Vita Ambria onlay
Other: IPs emax onaly — onlay restoration will be fabricated from lithium disilicate glass ceramic(IPS emax)
  Arms: IPS emax onlay

SUMMARY:
The 1ry objective will be to evaluate the amount of wear of onlays restorations made from VITA AMBRIA & IPS e.max Press and their opposing natural teeth.

2. The 2ry objective of the clinical trial will be to evaluate the fractures, retention, contact points, food impaction and radiographic examination of the VITA AMBRIA onlays compared with IPS e.max press onlays as defined by FDI criteria.

DETAILED DESCRIPTION:
A randomized controlled clinical trial, a double-blind (patient and examiner) is conducted by one trained and calibrated operators who perform all restorative procedures. The restorations are evaluated by a blind and calibrated two examiner using the FDI World Dental Federation criteria. A total of 24 patients will be randomly assigned to each group for a total of 48 patients. The randomization sequence will be generated (www.randomlists.com/team-generator) and to ensure the confidentiality of the allocation, this will be used opaque, sealed and numbered envelopes in series. These will be kept with an independent researcher for the moment of inclusion of the subjects.

Both groups will receive Onlay preparation . Digital impression by intra oral scanner will be taken, wax pattern for the onlay restoration will be designed and milled using CAD/CAM software. After that, the wax pattern will be invested and final onlay restoration will be constructed from VITA AMBRIA and IPS e.max press ingots according to manufacturing instructions. Primary outcome: The amount of wear will be evaluated according to FDI standard.

ELIGIBILITY:
Inclusion Criteria:

* The patient is healthy.
* 18-50 years old.
* Normal occlusion.
* Good oral hygiene.
* Tooth with complete root apex.
* Tooth with moderate coronal decay.

Exclusion Criteria:

• Patient Incapable of self-care, mental illness, undergoing radiotherapy, diabetic patient, allergy to one of the materials used, pregnancy, smoker, parafunctional habits, poor oral hygiene, severe periodontitis, tooth need vital pulp therapy or surgical crown lengthening or marginal elevation, tooth with enamel or dentin hypoplasia or hypocalcification, Mallaligned or malformed teeth and adjacent or opposing teeth are missed.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Wear evaluation | 1 year follow up
  The amount of wear will be defined as follows:
  1. Intra oral scanner will be used to scan the surface of the restorations and opposing natural enamel after achieving a complete dry surface by isolation.
  2. The recordings that measured at base line and 12 month periods will be superimposed on each other by specific software.
  3. Mean values and standard deviations of the amount of wear for all restorations' and opposing enamel's will be statistically analyzed.

SECONDARY OUTCOMES:
contact points and food impaction | 1 year follow up
  contact points and food impaction of the onlay restoration will be evaluated according to FDI standard (Grade 1-5), which has been defined as follows: Grade 1: Normal contact point (floss or 25 µm metal blade of can be inserted but not 50 µm blade).
  Grade 2: Slightly too strong but no disadvantage:
  Grade 3: Slightly too weak, no indication of damage to tooth, gingivae or periodontal structures (50 µm metal blade can pass easily but not 100 µm).
  Grade 4:Too weak (100 µm metal blade can pass) and possible damage (food impaction). Repair possible.
  Grade 5:Too weak and/or clear damage (food impaction) and/or pain/gingivitis. Requires replacement.
Radiographic examination | 1 year follow up
  Radiographic examination will be evaluated according to FDI standard (Grade 1-5), which has been defined as follows:
  Grade 1: No pathology, harmonious transition between restoration and tooth. Grade 2: (2.1) acceptable cement excess present ,(2.2) Positive/negative step present at margin<150 µm.
  Grade 3: (3.1) Marginal gap < 200 µm, (3.2)Negative steps visible < 250 µm and no adverse effects noticed,(3.3) Poor radiopacity of restorative material.
  Grade 4: (4.1) Marginal gap >250 µm, (4.2) Cement excess accessible but not removable,(4.3) Negative steps >250µm and repairable.
  Grade 5:(5.1) Secondary caries, large gaps ,(5.2) Apical pathology ,(5.3) Fracture/loss of restoration or tooth

CONTACTS AND LOCATIONS:
Overall Officials: Hussien RA Mohamed, Ph.D.Sc, Study Director — Assistant Professor of Crown and Bridge, Faculty of Dental Medicine, Al-Azhar University; Tamer AB Hamza, Professor, Study Chair — Professor of Crown and Bridge, Faculty of Dental Medicine, Al-Azhar University
Locations (1):
- Faculty of Dental Medicine , Al Azhar University, Cairo, Egypt

REFERENCES:
- [Background] Griffis E, Abd Alraheam I, Boushell L, Donovan T, Fasbinder D, Sulaiman TA. Tooth-cusp preservation with lithium disilicate onlay restorations: A fatigue resistance study. J Esthet Restor Dent. 2022 Apr;34(3):512-518. doi: 10.1111/jerd.12666. Epub 2020 Oct 3. PMID 33009726
- [Background] Lee JH, Myagmar G, Kwon HB, Han JS. A digital method for wear volume loss analysis using a single-scan three-dimensional dataset. J Dent Sci. 2022 Jan;17(1):638-641. doi: 10.1016/j.jds.2021.06.015. Epub 2021 Jul 4. PMID 35028110